CLINICAL TRIAL: NCT06844149
Title: Effects of a Cardiac and Psychosocial Rehabilitation Program on Depression, Anxiety, Self-Efficacy, Quality of Life, and Exercise Capacity in Young Adults With Fontan Circulation: A Randomized Controlled Trial
Brief Title: Impact of a Cardiac and Mental Health Rehab Program on Well-Being and Fitness in Young Adults With Fontan Circulation: A Randomized Trial
Acronym: (NCTXXXXXXXX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, June Huh, Professor of Pediatric Cardiology, Samsung Medical Center, Sungkyunkwan University School of Medicine, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-08-035---3; KCT0006496 (Registry Identifier: https://cris.nih.go.kr/)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiopulmonary Resuscitation; Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment model in which participants were randomly assigned to one of three groups: (1) a combined Cardiac and Psychosocial Rehabilitation (CPR) group, (2) a Cardiac Rehabilitation (CR) only group, or (3) a usual care control group. Each group received its assigned intervention throughout the study without crossover
Masking Description: "Not Applicable - This is an open-label study."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPR group; Cardiac and Psychosocial Rehabilitation (Experimental): Cognitive Behavioral Therapy (CBT)-based psychosocial rehabilitation program with a structured Home-Based Cardiac Rehabilitation (CR) program
  Interventions: Behavioral: CPR; (Cardiac and Psychosocial Rehabilitation) with Cardiac Rehabilitation
- CR group; Home-Based Cardiac Rehabilitation (Experimental): 8-week Home-Based Cardiac Rehabilitation (CR) program
  Interventions: Behavioral: CR; Home-Based Cardiac Rehabilitation
- Control group; usual care (Experimental): control group received usual care without any additional interventions
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: CPR; (Cardiac and Psychosocial Rehabilitation) with Cardiac Rehabilitation — This intervention combines an 8-week Cognitive Behavioral Therapy (CBT)-based psychosocial rehabilitation program with a structured Home-Based Cardiac Rehabilitation (CR) program for young adults with Fontan circulation. The CBT component includes weekly 90-minute group sessions focusing on stress management, cognitive restructuring, and social coping skills. The CR component consists of a personalized aerobic exercise plan, starting at 15-30 minutes per session and progressing to 40-60 minutes, with weekly monitoring and adjustments. This combined intervention is provided exclusively to participants in the CPR group
  Arms: CPR group; Cardiac and Psychosocial Rehabilitation
Behavioral: CR; Home-Based Cardiac Rehabilitation — This intervention consists of an 8-week Home-Based Cardiac Rehabilitation (CR) program designed for young adults with Fontan circulation. Participants follow a structured aerobic exercise plan tailored to their cardiopulmonary fitness levels. The program starts with 15-30 minutes of exercise per session, progressing to 40-60 minutes, with intensity set at 60-70% of maximum heart rate. Exercise adherence is monitored through weekly follow-ups, with adjustments made as needed. This intervention is provided to participants in both the CR group and the CPR group but without the Cognitive Behavioral Therapy (CBT) component in the CR-only group.
  Arms: CR group; Home-Based Cardiac Rehabilitation
Behavioral: Usual Care — Participants in the control group received usual care without any additional interventions. They did not participate in the Cognitive Behavioral Therapy (CBT)-Based Psychosocial Rehabilitation or the Home-Based Cardiac Rehabilitation (CR) programs during the study period. After the study was completed, they were given the option to enroll in the CPR program. This group serves as a comparison to evaluate the effectiveness of the interventions in the CPR and CR groups
  Arms: Control group; usual care

SUMMARY:
Helping Young Adults With Fontan Circulation Feel Better and Stay Active What is the study about? This study looked at how a special program could help young adults with Fontan circulation feel better mentally and physically. People with this condition often struggle with anxiety, depression, and low energy. The study tested a Cardiac and Psychosocial Rehabilitation (CPR) program, which included counseling and exercise training to improve their well-being.

Who participated?

38 young adults (ages 18-23) with Fontan circulation

They were divided into three groups:

CPR Group - received counseling (Cognitive Behavioral Therapy, CBT) and a home exercise program CR Group - did only the home exercise program Control Group - continued with their usual care What did the study find?

* Less anxiety and depression - The CPR group had the biggest improvement in mental health.
* Better self-confidence (self-efficacy) - Participants felt more capable of handling challenges.
* Higher quality of life - They felt happier and more engaged in daily life. ❌ No major changes in exercise ability - While they became more active, their heart fitness levels did not change much.

What does this mean for patients and families?

Mental health support is just as important as physical care for young adults with Fontan circulation.

A combination of counseling and exercise is better than exercise alone for reducing stress and anxiety.

Regular safe exercise should still be encouraged for better long-term health.

For healthcare providers:

This study supports adding psychological care (CBT) to standard cardiac rehabilitation.

More research is needed to optimize home-based exercise programs for Fontan patients.

Final message:

If you or a loved one has Fontan circulation, taking care of mental health is just as important as heart health. A program that includes counseling and exercise may help improve both!

DETAILED DESCRIPTION:
"All relevant information has been entered in the appropriate sections of the study record."

This ensures there is no unnecessary duplication while keeping the record clear and organized.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 23 years more than one year after Fontan surgery
* Had no surgery planned during study participation
* Had scores ≥ 8 for the anxiety (HADS-A) and/or depression (HADS-D) HADS subscales (Bjelland, Dahl, Haug, & Neckelmann, 2002; Holdgaard et al., 2023).
* Could read and complete the consent form and questionnaire, and participate in a Korean-language group

Exclusion Criteria:

* Undergoing psychotherapy during study participation
* Had significant cognitive impairment, psychosis, or personality disorder noted in their medical record
* Had scores ≥ 11 for HADS-D and > 17 for the Beck Depression Inventory (BDI) as evaluated by a psychiatrist or had been identified with severe depression or other serious psychiatric diagnoses (Kovacs et al., 2022; Marquez et al., 2020).
* Exhibited indications for the restriction of exercise of greater-than-moderate intensity based on recommendations from the American Heart Association (Franklin et al., 2020; Longmuir et al., 2013)

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Change in Depression Score Assessed by the Hospital Anxiety and Depression Scale (HADS- | Baseline, Week 8 (Post-Intervention), Week 12 (Follow-Up)
  Depression will be measured using the Hospital Anxiety and Depression Scale - Depression subscale (HADS-D). The HADS-D consists of 7 items, each scored from 0 to 3, with a total score ranging from 0 to 21. Higher scores indicate greater depressive symptoms. The primary outcome will be assessed at three time points: pre-intervention, post-intervention (week 8), and follow-up (week 12)

SECONDARY OUTCOMES:
Change in Anxiety Score Assessed by the Hospital Anxiety and Depression Scale (HADS-A) | Baseline, Week 8 (Post-Intervention), Week 12 (Follow-Up)
  Anxiety will be measured using the Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A). The HADS-A consists of 7 items, each scored from 0 to 3, with a total score ranging from 0 to 21. Higher scores indicate greater anxiety symptoms.
Change in Self-Efficacy Score Assessed by the General Self-Efficacy Scale (GSE) | Baseline, Week 8 (Post-Intervention), Week 12 (Follow-Up)
  Self-efficacy will be measured using the General Self-Efficacy Scale (GSE), a validated 10-item questionnaire scored on a scale from 1 to 4, with a total possible score of 10 to 40. Higher scores indicate greater self-efficacy.
Change in Quality of Life Score Assessed by the Linear Analog Scale (LAS) | Baseline, Week 8 (Post-Intervention), Week 12 (Follow-Up)
  Quality of life (QOL) will be measured using the Linear Analog Scale (LAS), a 10-cm visual analog scale ranging from 0 (worst) to 100 (best).
Change in Exercise Capacity Assessed by Cardiopulmonary Exercise Testing (CPET) | Baseline, Week 8 (Post-Intervention), Week 12 (Follow-Up)
  Exercise capacity will be measured using Cardiopulmonary Exercise Testing (CPET), assessing maximal oxygen uptake (VO₂ max), exercise duration, and metabolic equivalents (METs).
Change in Physical Activity Level Assessed by the International Physical Activity Questionnaire (IPAQ) Short Form | Baseline, Week 8 (Post-Intervention), Week 12 (Follow-Up)
  Physical activity (PA) was measured using the International Physical Activity Questionnaire (IPAQ) short form. The IPAQ categorizes PA levels as vigorous, moderate, or walking and quantifies total activity in metabolic equivalent of task minutes per week (MET-min/week).
Change in Heart Rate Variability (HRV) Assessed by Electrocardiographic Monitoring | Baseline, Week 8 (Post-Intervention), Week 12 (Follow-Up)
  Heart rate variability (HRV) was assessed using electrocardiographic (ECG) monitoring. HRV parameters include time-domain (e.g., standard deviation of NN intervals [SDNN], root mean square of successive differences [RMSSD]) and frequency-domain measures (e.g., low-frequency [LF], high-frequency [HF] power). Higher HRV indicates better autonomic function and cardiovascular health.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, 서울 - Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes will be shared upon reasonable request. Researchers can request access to the data by contacting the Principal Investigator